CLINICAL TRIAL: NCT02222506
Title: A Prospective Case Series Evaluating the Safety of the KLOX BioPhotonic System in Diabetic Foot Ulcers
Brief Title: Safety Evaluation of the KLOX BioPhotonic System in Diabetic Foot Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KLOX Technologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL-K1002-P009
Record Dates: First submitted 2014-08-19; First posted 2014-08-21 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-09

CONDITIONS: Diabetic Foot Ulcers
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- KLOX BioPhotonic System (Experimental): Treatment with KLOX BioPhotonic System in adjunction to Standard Of Care for diabetic foot ulcers.
  Interventions: Device: KLOX BioPhotonic System

INTERVENTIONS:
Device: KLOX BioPhotonic System — KLOX BioPhotonic System (Multi-LED Light and KLOX Photo Converter Wound Gel) will be administered until wound closure or for a maximum of 24 weeks, followed by a 8-week follow-up period, in association with Standard Of Care for diabetic foot ulcers.

SUMMARY:
The primary objective of these case series is to evaluate the safety and tolerability of the KLOX BioPhotonic System as adjunctive therapy to Standard Of Care (SOC) in patients with diabetic foot ulcers.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years of age and older;
* The subject or legal guardian must have signed an informed consent form;
* Female of child bearing potential must have a negative pregnancy test result at Baseline and both male and female patients must be willing to adhere to a medically-accepted birth control method during the course of the study;
* Willingness to return for all study visits;
* Willing and able to adhere to an off-loading protocol. Patient must adhere to wearing orthopedic shoe for the study duration (from first day of Screening until end of study);
* Target cutaneous, full thickness ulcer with University of Texas classification I-A (superficial, non-infected, non-ischemic wound not involving tendon, capsules, or bone) or II-A (non-infected, non-ischemic wound penetrating to tendon or capsule but not in the bone or joint). A patient with more than one diabetic foot ulcer may be included in the trial but only one ulcer will be selected for the investigational treatment, based on investigator's judgment;
* Ulcer present for more than 4 weeks prior to study entry (Screening/Visit 1);
* Ulcer area between 1 and 16 cm2 inclusive. The maximum diameter of the wound must not exceed 8 cm;
* Diabetes mellitus (Type 1 or 2) with an A1C < 12% at Screening;
* Diagnosis of neuropathic foot ulcer (10 grams pressure using Semmes-Weinstein 5.07 monofilament in the peri-ulcer area and/or biothesiometry or tuning fork 128 Hz);
* Wound area has not changed by more than +/- 30% between Screening visit and Week 1/Visit 1 (before treatment).
* Adequate arterial blood perfusion (ABI (ankle brachial index) between 0.7 and 1.3, inclusive, or toe pressure > 50 mmHg, or tcPO2 > 40 mmHg).

Exclusion Criteria:

* Diabetic foot ulcer present for more than 12 months;
* Target ulcer is over a deformity (such as Charcot deformity) that interferes with off-loading based on investigator's opinion;
* Patient cannot tolerate off-loading method;
* The ulcer to be treated is planned for operative debridement;
* The ulcer has significant necrotic tissue (e.g., more than 20% of the ulcer area);
* Major uncontrolled medical disorder(s) such as serious cardiovascular, renal, liver or pulmonary disease, lupus, palliative care or sickle cell anemia;
* Severe or significant hypoalbuminemia (albuminemia < 30 g/L, and/or pre-albumin < 5 mg/dL), or hypoproteinemia (proteinemia < 55g/L);
* Patient with moderate to severe anemia (Hb < 90g/L);
* Patient currently treated for an active malignant disease;
* Patient with history of malignancy within the wound;
* Patient with history of radiation therapy to the wound region;
* Patient with prior diagnosis of active malignant disease who is less than 1 year disease-free;
* Patient with a known osteomyelitis or active cellulitis;
* Patients that are immunosuppressed or on high dose chronic steroid use;
* Patients on systemic corticosteroids (a completion of corticosteroid course at least 30 days prior to study enrolment is required);
* Patient with active or systemic infection (note that the patient is however eligible for re-screening after the systemic infection has subsided);
* Successful revascularization surgery of the leg with the ulcer to be treated less than 8 weeks prior to Screening;
* Patients with severely uncontrolled diabetes mellitus (defined as A1C > 12%);
* Raynaud disease or other severe peripheral microvascular disease;
* Dermatologic comorbid disease (e.g., cutis laxa or collagen vascular disease);
* Active bleeding;
* Pregnancy, or breast feeding;
* Patients with bleeding diathesis;
* Patients on Warfarin or IV Heparin;
* The subject has any physical or psychiatric condition that in the Investigator's opinion would warrant exclusion from the study or prevent the subject from completing the study (e.g., severe morbid obesity, recent hip fracture, suspected non-compliance, etc.);
* Patients with ulcers from burns (from exposure to high heat), pressure ulcers or venous leg ulcers;
* Concurrent disease or drugs known to induce severe photosensitivity of the skin, such as porphyria;
* Patient has received biological-based therapy in any wound within 3 months of Screening;
* Concurrent participation in another clinical trial that involves an investigational drug or device that wound interfere with this study;
* Previous participation in other interventional wound healing clinical investigation within the 60 days prior to Screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-04; Primary Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of the KLOX BioPhotonic System in patients with diabetic foot ulcers. | 32 weeks
  Occurrence of adverse events, serious adverse events and incidents; pain assessment with Visual Analog Scale; clinical laboratory parameters; vital signs; physical examination; percentage of patients with clinical infection requiring systemic antimicrobial therapy; concomitant medications and treatments.

SECONDARY OUTCOMES:
Optimal frequency of treatment with KLOX BioPhotonic System on diabetic foot ulcers. | 32 weeks
  Exploration of the optimal frequency of treatment with KLOX BioPhotonic System on diabetic foot ulcers, with dosing flexibility according to Investigator's clinical opinion.
Rate of complete wound closure. | 32 weeks
Time to complete wound closure. | 32 weeks
Incidence of wound breakdown. | 32 weeks
Wound area reduction over time. | 32 weeks
Wound volume reduction over time. | 32 weeks

OTHER OUTCOMES:
Impact of treatment on Health-related quality of life. | 32 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Nikolis, Dr, Principal Investigator — Victoria Park MediSpa
Locations (3):
- Canada (3):
  - Q&T Research Chicoutimi, Chicoutimi, Quebec
  - Centre de Recherche Clinique de Laval, Laval, Quebec
  - Victoria Park MediSpa, Westmount, Quebec